CLINICAL TRIAL: NCT05076773
Title: A Comparative Study Between Ultrasound-guided Thoracic Paravertebral Block, Pectoral Nerves Block, and Erector Spinae Block for Pain Management in Cancer Breast Surgeries. A Randomized Controlled Study
Brief Title: TPVB, PECSB, ESPB for Postmastectmy Pain
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, kareem Mikhamer, Assistant fellow, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 32900654326
Record Dates: First submitted 2021-09-14; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (D) (Placebo Comparator): Patient will receive opioid only for management of their perioperative pain
  Interventions: Drug: IV morphine
- Paravertebral block Group (A) (Active Comparator): Will receive thoracic paravertebral block
  Interventions: Procedure: Ultrasound guided block; Drug: IV morphine
- Pectoral block Group (B) (Active Comparator): Will receive pectoral 1 and 2 block
  Interventions: Procedure: Ultrasound guided block; Drug: IV morphine
- Erector spinae block Group (C) (Active Comparator): Will receive erector spinae block
  Interventions: Procedure: Ultrasound guided block; Drug: IV morphine

INTERVENTIONS:
Procedure: Ultrasound guided block — Giving one regional block
  Other Names: Us guided paravertebral block; Us guided erector spinae block; Us guided PECs 1 and 2
  Arms: Erector spinae block Group (C); Paravertebral block Group (A); Pectoral block Group (B)
Drug: IV morphine — given when VAS>3

SUMMARY:
Aim of the work The aim of the study is to compare between the effects of ultrasound guided thoracic paravertebral block, pectoral nerve block II, and erector spinae block in management of pain during cancer breast surgeries. The hypothesis of the study is that the three groups will give comparative results.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status classification class I or II
2. Age group 18 - 60 years of the female gender
3. Patients undergoing breast cancer surgeries

Exclusion Criteria:

1. Patient refusal
2. History of hypersensitivity to local anesthetics
3. Bleeding disorders or patients receiving anticoagulants
4. Spine or chest wall deformities
5. Pregnancy
6. Local infection at the site of injection.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the study will be duration of analgesia (time to first rescue analgesia after administration of the block). | 0-24o minutess
  minutes

SECONDARY OUTCOMES:
Postoperative pain | 48 hours
  assessed by VAS score (0-10) where 0=no pain and 10=worst pain
Total morphine consumption | 48 hours
  recorded postoperatively in mg
Postoperative nausea and vomiting (PONV) | 48 hours
  4 points score of PONV (0-3) where 0=no PONV and 3=vomiting more than once

CONTACTS AND LOCATIONS:
Overall Officials: kareem M mikhimer, m.sc, Principal Investigator — assistant fellow, Ahmed Maher Hospital
Locations (1):
- Faculty of Medicine Menofia University, Shibīn al Kawm, Menofia, Egypt

IPD SHARING:
Plan to Share IPD: No
Title only